CLINICAL TRIAL: NCT07057882
Title: The Effect of Education Given to International University Students in Line With the HBM on Health Perception and Risky Behaviors: A Randomized Controlled Study
Brief Title: The Effect of Education Given to International University Students in Line With the Health Belief Model on Health Perception and Risky Behaviors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SakaryaU-HBMIntlEdu-RCT2025
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Health Behaviour; Risk Behavior, Health
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): "Participants will receive a Health Belief Model-based training program designed to improve health perception and reduce risky behaviors.".
  Interventions: Behavioral: Health Belief Model-based Education
- Control Group (No Intervention): "Participants will not receive any educational intervention during the study period."

INTERVENTIONS:
Behavioral: Health Belief Model-based Education — The intervention is a structured educational program based on the Health Belief Model (HBM), developed to improve health perception and reduce risky behaviors among international university students. The program includes six weekly sessions lasting approximately 45 minutes each, delivered face-to-face in small groups. The training content is tailored to address perceived susceptibility, severity, benefits, barriers, and self-efficacy related to health behaviors. Interactive discussions, visual materials, and culturally sensitive examples are used. Participants in the intervention group receive this training in addition to usual care or routine university services..
  Arms: Intervention Group

SUMMARY:
The World Health Organization defines health as a state of complete physical, mental, and social well-being. Health is a process in which individuals adapt to environmental changes, and this process is influenced by beliefs, experiences, and health behaviors. Health perception is a combination of an individual's thoughts about their own health and is a significant indicator of both physical and mental well-being. University students enter a new phase of life that can affect their health perceptions, during which they may experience health problems associated with factors such as stress, physical activity, and nutrition. International students, in particular, may encounter additional challenges during the cultural adaptation process and may engage in risky behaviors that affect their health behaviors.The Health Belief Model (HBM) is a framework used to understand and modify individuals' health behaviors. This study examines the effectiveness of an HBM-based educational intervention in evaluating international students' health perceptions and risky behaviors. While the literature supports the effectiveness of HBM-based education in reducing risky behaviors, there is a lack of randomized controlled trials conducted specifically with international students.This study, to be conducted with international students at Sakarya University, aims to improve students' health perceptions and reduce risky behaviors. The research is designed as a randomized controlled trial with pre-test/post-test, single-blind, experimental and control groups. It is expected that the HBM-based educational intervention delivered to the experimental group will enhance international university students' health perceptions and reduce their likelihood of engaging in risky behaviors.Data collection tools include the "Health Perception Scale" and the "Risky Behaviors Scale - University Form". Data obtained in the study will be analyzed using the SPSS (Statistical Package for the Social Sciences) for Windows 22.0 software.

ELIGIBILITY:
Inclusion Criteria:- To study at Sakarya University as an international student

* To have passed the Turkish language proficiency (speaking Turkish at C1 level)
* Volunteering and giving consent to participate in the research
* Being open to communication and cooperation
* No diagnosed psychiatric illness
* Scoring below the average scale score of the sample group for the "Health Perception Scale" and above the average scale score of the sample group for each sub-dimension of the "Risky Behaviors Scale University Form" scale-

Exclusion Criteria:- To study at Sakarya University as an international student

* To have passed the Turkish language proficiency (speaking Turkish at C1 level)
* Volunteering and giving consent to participate in the research
* Being open to communication and cooperation
* No diagnosed psychiatric illness
* Scoring below the average scale score of the sample group for the "Health Perception Scale" and above the average scale score of the sample group for each sub-dimension of the "Risky Behaviors Scale University Form" scale

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
change in health perception and risky behaviors scores | Baseline and one month and three months after intervention
  Measured using the Perception of Health Scale and University Form of Risk Behavaiors Scale comparing pre- and post-intervention scores among international students. The lowest and highest scores that can be obtained from the Health Perception Scale are 15 and 75, respectively. A high total score indicates high health perceptions and a low total score indicates low health perceptions.Since the dimensions of the Risky Behaviors Scale University Form are not interrelated, the scale does not give a total score, and the scores obtained from each dimension are evaluated separately. However, the scale does not have a cut-off score and a high score in each dimension indicates a higher level of risk in that dimension.

IPD SHARING:
Plan to Share IPD: No